CLINICAL TRIAL: NCT02148562
Title: Assessment of Hepatitis B Virus Intra-host Population and Host-specific Immune Marker Diversity With Next-generation Sequencing: From Chronic Infection to End-stage Liver Disease and Liver Cancer
Brief Title: Assessment of Hepatitis B Virus Intra-host Population and Host-specific Immune Marker Diversity
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Fund for Scientific Research, Flanders, Belgium (Other)
Responsible Party: Principal Investigator, MahmoudReza Pourkarim, PhD, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S56121; 12G1714N (Other Grant/Funding Number: Fund for Scientific Research Flanders)
Record Dates: First submitted 2014-04-04; First posted 2014-05-28 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Hepatitis B; Hepatitis B, Chronic; End Stage Liver Disease; Carcinoma, Hepatocellular
MeSH Terms: conditions — Hepatitis B; Hepatitis B, Chronic; End Stage Liver Disease; Carcinoma, Hepatocellular

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Chronic Hepatitis B: Diagnosis of Hepatitis B related liver disease in a pre-advanced stage
- End stage liver disease: Diagnosis of advanced liver disease related to Hepatitis B

SUMMARY:
In this project proposal, the investigators will investigate the genetic alterations of Hepatitis B Virus (HBV) strains circulating in Belgian patients who developed end stage liver disease. Additionally, the investigators will compare and link these data sets with three genetic factors involved in immune system response.

DETAILED DESCRIPTION:
This project proposes to identify and characterize the genetic alterations associated with intra-host evolution of HBV from a chronically infection status to an end-stage liver disease status.

ELIGIBILITY:
Inclusion Criteria:

Study group:

* Clinical diagnosis of advanced liver disease related to chronic Hepatitis B infection (cirrhosis, hepatocellular carcinoma,..)
* Availability of serum samples

Control group:

* Clinical diagnosis of liver disease related to chronic Hepatitis B infection in a pre-advanced stage
* Matched demographic and geographic characteristics to study group
* Availability of serum samples

Exclusion Criteria:

* Liver disease caused by other hepato-tropic viruses
* Patients with auto-immune diseases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with liver disease related to Hepatitis B in a pre-advanced (chronic infection) and advanced stage (end-stage liver diseases) treated at the Hepatology Department of University Hospital of Leuven
Sampling Method: Non-Probability Sample
Enrollment: 274 (Estimated)
Dates: Start 2014-04; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
genetic variants of Hepatitis B | 6 months
  Virus variants will be identified by amino acid or nucleotide variations (insertions or deletions) in different Open Readind Frames (ORFs) of the HBV genome by using next-generation sequencing.
  Comparison of virus variants within one patient Comparison of virus variants between patients with end stage liver disease and patients with a chronic Hepatitis B infection.
  Determination of the viral load by quantitative Polymerase Chain Reaction (PCR).

SECONDARY OUTCOMES:
genetic variation in host-specific immune markers | at day of enrollment
  Amplification of HLA-A, HLA-B, HLA-C class I and HLA class II using PCR methods and next-generation sequencing
  Amplification of KIR genes: 2DS1, 2DS2, 2DS3, 2DS4, 2DS5, 3DS1 and 1D, 2DL1 2DL2, 2DL3, 2DL5 and 3DL1 using PCR methods and next-generation sequencing
  Amplification of SNPs in TNF alfa, TGF beta1 and IFN-R using PCR methods and next-generation sequencing

CONTACTS AND LOCATIONS:
Overall Officials: MahmoudReza Pourkarim, PhD, Principal Investigator — UZ Leuven campus Gasthuisberg, Herestraat 49. 3000 Leuven, Belgium
Locations (1):
- University Hospitals Leuven campus Gasthuisberg, Leuven, Flemish Brabant, Belgium